CLINICAL TRIAL: NCT03602846
Title: Diabetes in Pregnancy, Therapy and Pregnancy Outcomes
Brief Title: Diabetes in Pregnancy and Pregnancy Outcomes
Status: Completed | Type: Observational
Sponsor: Tarumanagara University (Other)
Collaborators: Hermina Podomoro Hospital (Unknown)
Responsible Party: Principal Investigator, Anthony Paulo Sunjaya, Principle Investigator, Tarumanagara University
Other Study IDs: APS002
Record Dates: First submitted 2018-06-27; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus in Pregnancy; Diabetes, Gestational
Keywords: diabetes mellitus in pregnancy; gestational diabetes; pregnancy outcomes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Nutrition Therapy; Insulin; Hypoglycemic Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Good Outcome: Good outcome is defined as the safe delivery of the newborn.
  Interventions: Dietary Supplement: Medical Nutrition Therapy; Drug: Insulin; Drug: Oral Antidiabetics
- Poor Outcome: Poor outcome is defined as the incidence of fetal demise during pregnancy.
  Interventions: Dietary Supplement: Medical Nutrition Therapy; Drug: Insulin; Drug: Oral Antidiabetics

INTERVENTIONS:
Dietary Supplement: Medical Nutrition Therapy — Only given medical nutrition therapy.
Drug: Insulin — Prescribed with rapid acting, intermediate acting, mixed or long acting insulin.
Drug: Oral Antidiabetics — Prescribed with all types of oral anti-diabetics.

SUMMARY:
To compare the clinical, glycemic profile and therapy as well as pregnancy complications and infant mortality among diabetic mothers in Indonesia.

DETAILED DESCRIPTION:
Pregnancy is a diabetogenic state with increasing burden on the mother's metabolism. Insulin resistance is often found during pregnancy leading to a compensatory increase in pancreatic β-cell response and eventually hyperinsulinemia. Undiagnosed and untreated diabetes in pregnancy have been shown to be linked with numerous comorbidities and complications to both mother and foetus.

This study aims to compare the clinical, glycemic profile along with comorbidities, management and outcomes of diabetic mothers. Pregnant mothers with gestational and pregestational diabetes diagnosed under the ICD-10 coding of O24 were included in this study. The inclusion criteria was all patients with primary diagnosis of O24, have visited the clinic at least twice with a complete record of glycemic profile, management and fetal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and laboratory diagnosis of Diabetes in Pregnancy (Gestational and Pregestational diabetes)
* Mothers must have visited the clinic at least twice throughout their pregnancy, at least one at the first trimester and one at the third trimester

Exclusion Criteria:

* Pregnancy is still undergoing
* Incomplete record of glycemic profile, management and fetal outcomes

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant mothers with gestational and pregestational diabetes diagnosed under the ICD-10 coding of O24.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Infant Mortality | Throughout the length of pregnancy, an average of 9 months
  Infant Mortality either due to abortion, intrauterine fetal death or stillbirth as recorded in medical records
Gestational Age at Birth | At time of delivery
  Infant Gestational at Birth as recorded in medical records
Infant Body Weight | At time of delivery
  Infant Body Weight as recorded in medical records
Infant Body Length | At time of delivery
  Infant Body Length as recorded in medical records
Infant Head Circumference | At time of delivery
  Infant Head Circumference as recorded in medical records
APGAR Score | At time of delivery
  One and five minute APGAR Scores as recorded in medical records

SECONDARY OUTCOMES:
Maternal Mortality | Throughout the length of pregnancy, an average of 9 months
  Maternal death as recorded in medical records
Comorbidities | Throughout the length of pregnancy, an average of 9 months
  Comorbid conditions were defined as either concomitant hypertension, anemia, urinary tract infection, preeclampsia/eclampsia, or combinations of them as recorded in medical records
Method of Delivery | At time of delivery
  Vaginal Birth or Caesarean Section as recorded in medical records

OTHER OUTCOMES:
Random Plasma Glucose | Throughout the length of pregnancy, an average of 9 months
  Random Plasma Glucose levels as recorded in medical records
Fasting Plasma Glucose | Throughout the length of pregnancy, an average of 9 months
  Fasting Plasma Glucose levels as recorded in medical records
Oral Glucose Tolerance Test | Throughout the length of pregnancy, an average of 9 months
  Oral Glucose Tolerance Test levels as recorded in medical records
Glycated Hemoglobin (HbA1c) | Throughout the length of pregnancy, an average of 9 months
  Glycated Hemoglobin (HbA1c) levels as recorded in medical records

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Sunjaya, Principal Investigator — Tarumanagara University

IPD SHARING:
Plan to Share IPD: Undecided